CLINICAL TRIAL: NCT01090336
Title: Prevalence of Inadequate Platelet Inhibition After Oral Loading With Prasugrel/Clopidogrel in Patients With an Acute Coronary Syndrome Undergoing Early PCI
Brief Title: Prasugrel Versus Clopidogrel in Acute Coronary Syndrome (ACS) Undergoing Percutaneous Coronary Intervention (PCI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Prof. Dr. Evangelos Giannitsis, Department of Cardiology, University of Heidelberg
Other Study IDs: PC01; S-235/2009 (Other: Ethics committee of the University of Heidelberg)
Record Dates: First submitted 2010-03-16; First posted 2010-03-19 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2010-03

CONDITIONS: Patients With Acute Coronary Syndrome
Keywords: platelet aggregation inhibition; prasugrel; clopidogrel; ACS

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clopidogrel group: At the discretion of the attending cardiologist patients are treated with clopidogrel (600mg loading and 75mg daily dose)
- Prasugrel group: At the discretion of the attending cardiologist patients are treated with prasugrel (60mg loading and 10mg daily dose)

SUMMARY:
Background: Both prasugrel and clopidogrel are prescribed drugs which compete as platelet inhibitors in patients with acute coronary syndrome (ACS). Whether rates of drug resistance/hyporesponsiveness are lower with prasugrel and whether more consistent and earlier onset of platelet inhibition may reduce infarct size in patients with ACS undergoing early PCI remains, at present, unknown.

Study design/study population: This trial is a prospective, open-label, single centre observational trial. Patients receive either prasugrel (60mg) or clopidogrel (600mg) at the discretion of the attending cardiologist. Patients with exclusion criteria for prasugrel will be excluded for clopidogrel as well. The study population includes 80 subjects with moderate to high-risk ACS, ie patients with unstable angina (UA) and non-ST-segment elevation MI (NSTEMI) and TIMI risk score of 3 or higher, within 72 hours after onset of symptoms. In all patients early PCI is planned.

Study objective/endpoint/methods: The primary objective of this trial is to evaluate whether rates of hyporesponsiveness are lower with prasugrel and whether more consistent and earlier onset of platelet inhibition may reduce infarct size in ACS in patients undergoing early PCI.

The primary endpoint is the rate of drug resistance at time of index intervention. Optical and impedance aggregometry using ADP (5 and 20 μM) and collagen (1 μg/ml) as platelet agonists is used to measure platelet aggregation. Addition of the specific antagonists aspirin and mesamp to the probe is used to discriminate between pharmacodynamic and pharmacokinetic drug resistance.

Secondary endpoint is the reduction of myocardial infarct size determined by post-interventional increase of high sensitive TnT (TnT hs) during the days following the index event reflecting earlier, more effective and more consistent inhibition of platelet function.

Tertiary endpoint is the composite clinical endpoint of cardiovascular death, nonfatal MI, or stroke and urgent target vessel revascularization during hospitalization and after 6 and 12 months.

Safety endpoint is any TIMI major or minor bleeding during hospital stay and after 6 and 12 months including intracranial and life-threatening bleeding.

DETAILED DESCRIPTION:
look above

ELIGIBILITY:
Inclusion criteria:

* Patients with unstable angina or non-ST-elevation myocardial infarction with ischemic symptoms lasting 10 minutes or more and occurring within 72 hours before randomization,
* A TIMI risk score of 3 or more, and
* Either ST-segment deviation of 1 mm or more or elevated levels of a cardiac biomarker of necrosis.
* Legal age (and ≥18 y) and competent mental condition to provide written informed consent

Exclusion Criteria:

* Patients with weight < 60 kg, age > 75 year or history of TIA, stroke or intracranial bleeding according to prasugrel contraindications
* Clinical status forbid inclusion (eg cardiogenic shock at the time of randomization, refractory ventricular arrhythmias, New York Heart Association class IV congestive heart failure etc)
* Bleeding risk exclusion criteria including fibrin-specific and non-fibrin-specific fibrinolytic therapy for index event, active internal bleeding or history of bleeding diathesis or any clinical findings in the judgment of the investigator associated with an increased risk of bleeding
* History of hemorrhagic stroke, intracranial neoplasm, arteriovenous malformation, or aneurysm
* Ischemic stroke within 3 months prior to screening
* Oral anticoagulation or INR greater than 1.5 at the time of screening
* Platelet count of less than 100 000/mm3 at the time of screening
* Anemia (hemoglobin <10 g/dL) at the time of screening
* Prior/concomitant therapy with thienopyridine or daily treatment with nonsteroidal antiinflammatory drugs or cyclooxygenase-2 inhibitors
* General exclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes 80 subjects with moderate to high-risk ACS, ie patients with unstable angina (UA) and non-ST-segment elevation MI (NSTEMI) and TIMI risk score of 3 or higher, within 72 hours after onset of symptoms. In all patients early PCI is planned. Patients with exclusion criteria for prasugrel will be excluded for clopidogrel as well.
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2009-08; Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the rate of drug resistance at time of index intervention. | Routinely, platelet aggregation is evaluated ideally daily up to 96 hours after index event.
  Platelet aggregation is determined by light transmission and impedance aggregometry as previoulsy described (Boris T. Ivandic, Philipp Schlick, Peter Staritz, Kerstin Kurz, Hugo A. Katus and Evangelos Giannitsis: Determination of Clopidogrel Resistance by Whole Blood Platelet Aggregometry and Inhibitors of the P2Y12 Receptor; Clinical Chemistry 52: 383-388, 2006)

SECONDARY OUTCOMES:
Secondary endpoint is the reduction of myocardial infarct size determined by post-interventional increase of high sensitive TnT (TnT hs). | Routinely, ideally daily until 96h after index event.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giannitsis, Prof. Dr., Principal Investigator — Department of Cardiology, University of Heidelberg
Locations (1):
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Ivandic BT, Schlick P, Staritz P, Kurz K, Katus HA, Giannitsis E. Determination of clopidogrel resistance by whole blood platelet aggregometry and inhibitors of the P2Y12 receptor. Clin Chem. 2006 Mar;52(3):383-8. doi: 10.1373/clinchem.2005.059535. Epub 2006 Jan 19. PMID 16423907